CLINICAL TRIAL: NCT00577356
Title: Phase II Trial of Neoadjuvant Docetaxel and CG1940/CG8711 Followed by Radical Prostatectomy in Patients With High-Risk, Clinically Localized Prostate Cancer
Brief Title: Docetaxel and Immunotherapy Prior to Prostatectomy for High-Risk Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety reasons, though no safety issues arose.
Sponsor: Benaroya Research Institute (Other)
Collaborators: Cell Genesys (Industry); Sanofi (Industry)
Responsible Party: Jacqueline Vuky, MD, Virginia Mason Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB07028; I-0057; IST# 16194
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Results first posted 2011-01-20 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2010-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 75mg/m2 will be given intravenously every 3 weeks for four cycles.
  Other Names: Taxotere
Biological: CG1940/CG8711 — Immunotherapy allogeneic GM-CSF secreting cellular vaccine

SUMMARY:
The purpose of this study is to find out what effects, good and bad, the combination of docetaxel with CG1940/CG8711 (immunotherapy drugs) have on destroying prostate cancer before removal the prostate (prostatectomy).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have clinical stage 1-3 disease and no radiographic evidence of metastatic disease
* Nomogram Prediction: Patients must have a Kattan nomogram predicted probability of being free from biochemical progression at 5 years after surgery of <60%.

Exclusion Criteria:

* Concurrent or prior treatment with radiation, cytotoxic or biologic therapy for prostate cancer, prior hormonal therapy (except finasteride or dutasteride for obstructive voiding symptoms)
* Male patients unwilling to use effective means of contraception are excluded. Contraception should be continued for 3 months after treatment.
* Prior malignancy will not exclude the patient. (Patients can not have active cancer or be undergoing active treatment). The Principal Investigator will make final decision regarding eligibility since the end point is pathological complete response.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Vuky, MD, Principal Investigator — Virginia Mason Medical Center
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States

REFERENCES:
- See also: Related Info — http://benaroyaresearch.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from Feb. 08 through September 08 at Virginia Mason Medical Center
Pre-assignment Details: Eligible patients had histologically confirmed adenocarcinoma of the prostate with clinical stage 1-3, no evidence of metastatic disease, and were appropriate candidates for radical prostatectomy with an estimated life expectancy >10 years.
Groups:
- CG1940/CG8711 (Immunotherapy Drug): Patients were given a prime immunotherapy of 5 x 108 cells consisting of equal amounts of CG1940 and CG8711 followed 21 days later by boost immunotherapies of 3 x 108 cells consisting of equal amounts of CG1940 and CG8711 every 21 days for the first 4 immunotherapies. (given 2 to 3 days after docetaxel) for a total of 4 immunotherapies, followed by a fifth dose given at 2, 8, or 14 days prior to prostatectomy, and then beginning at 3 - 6 weeks post-operatively an additional 6 immunotherapies every 14 days for a combined total of 11 immunotherapies. Docetaxel chemotherapy was administered intravenously starting day 1 of the first week and given every 3 weeks thereafter for a total of 4 cycles. A cycle is defined as every 21 days (3 weeks).
Period: Overall Study
Arm/Group | CG1940/CG8711 (Immunotherapy Drug)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CG1940/CG8711 (Immunotherapy Drug)
Number analyzed (Participants) | 6
Age, Customized [Number; unit: participants]
  <55 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 6
adenocarcinoma of the prostate and no radiographic evidence of metastatic disease [Mean (Standard Deviation); unit: years] | 2 (7.1)
Prostate Cancer [Number; unit: participants] | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pathological Complete Response.
Description: CG1940/CG8711 was given along with docetaxel over a series of treatment prior to radical prostatectomy. Pathology of resected specimen was done to determine complete response, defined as no microscopic evidence of neoplastic cells in the resected specimen
Time Frame: The study evaluates 4 months of docetaxel and immunotherapy prior to radical prostatectomy followed by radical prostatectomy with an additional 3 months of immunotherapy after radical prostatectomy.
Population: Study was stopped before analysis occured.
Measure: Number; unit: participants
Arm/Group | CG1940/CG8711 (Immunotherapy Drug)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | CG1940/CG8711 (Immunotherapy Drug)
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
the trial was closed prior to planned accrual of 30 patients due to an external report from the randomized trial of docetaxel and CG1940/CG8711 resulting in a higher incidence of deaths compared to docetaxel alone in metastatic prostate cancer.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No